CLINICAL TRIAL: NCT05163093
Title: Research on the Diagnosis and Treatment of Angle Closure Glaucoma With Abnormal Lens Zonular
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chunyan Qiao_2021 (Other)
Responsible Party: Sponsor-Investigator, Chunyan Qiao_2021, Ophthalmologist, Chief of out-patient department, Beijing Tongren Hospital
Organization: Beijing Tongren Hospital (Other)
Other Study IDs: Angle closure glaucoma
Record Dates: First submitted 2021-11-07; First posted 2021-12-20 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Angle-Closure Glaucoma
Keywords: angle closure glaucoma; lens subluxation; zonular
MeSH Terms: conditions — Glaucoma, Angle-Closure; Lens Subluxation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lens capsule
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Angle closure glaucoma patients with or without abnormal zonular.: We observe the zonular during surgery, and divide patients into two groups according to their zonular, including with or without abnormal zonular.
- Patients with age-related cataract.: We observe the zonular during surgery, and divide patients into two groups according to their zonular, including with or without abnormal zonular.

SUMMARY:
Angle-closure glaucoma is the main type of glaucoma in China, which is divided into acute and chronic angle-closure glaucoma. Previous studies from our group have found that, in lens excision combined with glaucoma surgery, accounted for 46.2% of patients were ligament abnormalities, such as lens subluxation with suspensory ligament relaxation. And it was more common in acute angle-closure glaucoma (55.8%). In acute angle-closure glaucoma, approximately 55.2% of suspensory ligament abnormalities were not diagnosed preoperatively depend on UBM and slit lamp examinations. The purpose of this study was to find a better preoperative diagnosis method of the suspensory ligament abnormality, and to observe the influence of the suspensory ligament abnormality on the occurrence, development and treatment effect of acute angle-closure glaucoma. We plan to collect patients with acute angle-closure glaucoma with monocular onset and exclude traumatic, secondary glaucoma and a history of intraocular surgery. The onset eyes were treated with combined operation, and divided into two groups according to the presence or absence of suspensory ligament abnormalities. The fellow eyes were treated with laser peripheral iridectomy, and followed examination, including UBM, anterior-segment OCT, and IOL master 700, before and after bow excitation test. Then follow up patients every six months. Ultimately, the fellow eyes will be treated with combined surgery after 2.5 years or the fellow eyes occur acute angle-closure glaucoma. In the end, we evaluate the sensitivity and specificity of each index, and the influence of suspensory ligament abnormality on angle-closure glaucoma progression.

DETAILED DESCRIPTION:
1.Inclusion criteria:

(1)age: 45-79 years old, BCVA>0.3, 19mm<axial length<24mm. (2).Continuous cases diagnose with angle-closure glaucoma in Beijing Tongren Hospital from January 1st, 2022 to December 31th, 2023 and undergo phacoemulsification lens extraction combined with intraocular lens implantation combined with anterior chamber angle separation will be included in the case group. (3). The patients who are diagnosed age-related cataract and undergo phacoemulsification lens extraction combined with intraocular lens implantation at the same time in Beijing Tongren Hospital will be included as control group. (4). All the surgeries were finished by the same two experienced ophthalmologists. (5). Both eyes will be undergo with surgery, and we will include the first eye for observation.

2.Exclusion critieria:

(1)Age-related cataract patients whose anterior chamber depth (ACD)<2.5mm, 22mm>axial length, or axial length>26mm. (2).Patients who underwent ocular surgery, such as peripheral iridotomy, trabeculectomy. (3). Patients with history of ocular trauma. (4).Patients with other ophthalmic diseases that can cause shallow anterior chamber expect glaucoma and cataract, such as choroid detachment, ciliary body detachment, retinal detachment, bulbar tumor, etc. (5). Secondary glaucoma, such as neovascular glaucoma.

3.Diagnostic critieria:

1. angle-closure glaucoma (ACG): a. Both eyes with shallow anterior chamber (ACD<2.5mm). b. With short axial length (axial length<24mm).
2. acute angle-closure glaucoma (AACG): a. Both eyes with ACG characteristic anatomical structure, including shallow anterior chamber and short axial length. b.Patients with classic history of acute episode, acute elevated intraocular pressure, and atrioscopy or ultrasound biomicroscope (UBM) examination indicated angle closure. c. Ocular examination showed the characteristic changes of acute ocular hypertension: iris atrophy, dilated pupil, glaucoma spot, and pigmented Kp.

4. Diagnostic criteria for lens suspensory ligament abnormalities

1. . Pre-operation: a. UBM shows the distance from ciliary processes to the equatorial part of lens varies in different directions. b. ACD are different between the two eyes and/or lens iris septum tremors by slit-lamp examination.
2. .Intraoperation: a. Suspensory ligament relaxation: with obvious radial folds on lens anterior capsules during continuous circular capsulorhexis (CCC), and could not observe the equator of lens. b. Rupture of suspensory ligament: could observe the equator of lens after full dilation of the pupil.

ELIGIBILITY:
Inclusion criteria:

1. age: 45-79 years old, BCVA>0.3.
2. Clinical diagnosis of angle-closure glaucoma, with 19mm<axial length<24mm.
3. Clinical diagnosis of age-related cataract (as control group), with 22mm<axial length<26mm.
4. All the surgeries were finished by the same two experienced ophthalmologists.
5. The first operated eye was included for observation.

Exclusion criteria:

1. Age-related cataract patients whose anterior chamber depth (ACD)<2.5mm.
2. Patients who underwent ocular surgery, such as peripheral iridotomy, trabeculectomy.
3. Patients with history of ocular trauma.
4. Patients with other ophthalmic diseases that can cause shallow anterior chamber expect glaucoma and cataract, such as choroid detachment, ciliary body detachment, retinal detachment, bulbar tumor, etc.
5. Secondary glaucoma, such as neovascular glaucoma.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous cases diagnose with angle-closure glaucoma in Beijing Tongren Hospital from January 1st, 2022 to December 31th, 2023 and undergo phacoemulsification lens extraction combined with intraocular lens implantation combined with anterior chamber angle separation will be included in the case group. And the patients who are diagnosed age-related cataract and undergo phacoemulsification lens extraction combined with intraocular lens implantation at the same time in Beijing Tongren Hospital will be included as control group.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
visual acuity (VA) | baseline
  best corrected visual acuity (BCVA)
visual acuity (VA) | during the procedure
  best corrected visual acuity (BCVA)
intraocular pressure (IOP) | baseline
  non-contact tenometer
intraocular pressure (IOP) | during the procedure
  non-contact tenometer
slit-lamp examination | baseline
  Assess the condition of ACD and lens iris septum tremors by slit-lamp examination
slit-lamp examination | during the procedure
  Assess the condition of ACD and lens iris septum tremors by slit-lamp examination
gonioscopy | baseline
  Observe the range of peripheral anaterior synechia by gonioscopy
gonioscopy | during the procedure
  Observe the range of peripheral anaterior synechia by gonioscopy
IOL Master 700 | baseline
  Assess the anterior chamber depth (ACD)
IOL Master 700 | baseline
  lens thickness (LT)
IOL Master 700 | baseline
  axial length (AL)
IOL Master 700 | baseline
  calculate lens position(LP). LP=ACD+1/2LT.
IOL Master 700 | baseline
  relative lens position. RLP=LP/AL.
IOL Master 700 | during the procedure (before bend test)
  Assess the anterior chamber depth (ACD)
IOL Master 700 | during the procedure (before bend test)
  lens thickness (LT)
IOL Master 700 | during the procedure (before bend test)
  axial length (AL)
IOL Master 700 | during the procedure (before bend test)
  calculate lens position(LP). LP=ACD+1／2LT.
IOL Master 700 | during the procedure (before bend test)
  relative lens position. RLP=LP/AL.
IOL Master 700 | during the procedure (after bend test)
  Assess the anterior chamber depth (ACD)
IOL Master 700 | during the procedure (after bend test)
  lens thickness (LT)
IOL Master 700 | during the procedure (after bend test)
  axial length (AL)
IOL Master 700 | during the procedure (after bend test)
  calculate lens position(LP). LP=ACD+1／2LT.
IOL Master 700 | during the procedure (after bend test)
  relative lens position. RLP=LP/AL.
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  Assess the ACD
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  angle opening distance (AOD)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  trabecular-iris space area (TISA)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  angle recess area (ARA)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  iris-trabecular index of contact (ITIC)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  Front R
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  Back R
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  Tilt
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  Lens thickness (LT)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  Decent
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  LE-Dia
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | baseline
  lens vault (LV)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  Assess the ACD
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  angle opening distance (AOD)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  trabecular-iris space area (TISA)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  angle recess area (ARA)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  iris-trabecular index of contact (ITIC)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  Front R
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  Back R
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  Tilt
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  Lens thickness (LT)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  Decent
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  LE-Dia
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (before bend test)
  lens vault (LV)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  Assess the ACD
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  angle opening distance (AOD)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  trabecular-iris space area (TISA)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  angle recess area (ARA)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  iris-trabecular index of contact (ITIC)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  Front R
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  Back R
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  Tilt
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  Lens thickness (LT)
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  Decent
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  LE-Dia
CAISA 2 anterior segment optical coherence tomography (AS-OCT) | during the procedure (after bend test)
  lens vault (LV)
Ultrasound biomicrospy (UBM) | baseline
  Measure the distance between ciliary and the equator of lens, iris-lens angle by using UBM. Collect all the data of 3, 6, 9,12 o'clock position.
Ultrasound biomicrospy (UBM) | during the procedure (before bend test)
  Measure the distance between ciliary and the equator of lens, iris-lens angle by using UBM. Collect all the data of 3, 6, 9,12 o'clock position.
Ultrasound biomicrospy (UBM) | during the procedure (after bend test)
  Measure the distance between ciliary and the equator of lens, iris-lens angle by using UBM. Collect all the data of 3, 6, 9,12 o'clock position.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China